CLINICAL TRIAL: NCT06664216
Title: Impact of Behavioral Compliance Between Residents and Surgeons Using a Simulation Environment of Trocar Placement in Laparoscopic Cholecystectomy
Brief Title: Impact of Behavioral Compliance Between Residents and Surgeons
Acronym: CONF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Excelencia en Enfermedades de Cabeza y Cuello (Other)
Collaborators: Asociacion Colombiana de Cirugia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3
Record Dates: First submitted 2024-08-04; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Conformity, Social
Keywords: conformity; groupthinking; surgeons
MeSH Terms: conditions — Social Conformity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants use a laparoscopic model without any previous marks.
  Interventions: Behavioral: incorrect trocar placement marks.
- Intervention (Experimental): Participants use a laparoscopic model with incorrect trocar placement marks.
  Interventions: Behavioral: incorrect trocar placement marks.

INTERVENTIONS:
Behavioral: incorrect trocar placement marks. — Participants in the experimental group will perform trocar placements on laparoscopic models that have been pre-marked with incorrect insertion sites by previous participants. These marks simulate procedural steps or anatomical landmarks that are intentionally incorrect.

SUMMARY:
This study aims to evaluate the influence of perceived peer performance on the clinical skill of trocar placement during laparoscopic cholecystectomy among surgeons and surgical residents. It investigates whether exposure to incorrect trocar placements by peers affects the accuracy of subsequent placements.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Spanish mother tongue
* Experience in laparoscopic cholecystectomy
* Consent to participate

Exclusion Criteria:

* Physical disability preventing understanding or response
* More than 3 years of suspension from surgical practice

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
accuracy of the trocar placements | 1 week
  The participant must define in a graphic format the site where the trocars would be placed to perform a laparoscopic cholecystectomy.
  The number of trocars correctly placed will be recorded. A rate of will be calculated: Trocars in the correct place/Total number of trocars.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociacion Colombiana de Cirugia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cialdini RB, Goldstein NJ. Social influence: compliance and conformity. Annu Rev Psychol. 2004;55:591-621. doi: 10.1146/annurev.psych.55.090902.142015. PMID 14744228
- [Result] MILGRAM S. BEHAVIORAL STUDY OF OBEDIENCE. J Abnorm Psychol. 1963 Oct;67:371-8. doi: 10.1037/h0040525. No abstract available. PMID 14049516
- [Result] Kass LR. Ethical dilemmas in the care of the ill. I. What is the physician's service? JAMA. 1980 Oct 17;244(16):1811-6. PMID 7420682
- [Result] Tobin B. Respect for conscientious judgement in health care. J Paediatr Child Health. 2022 Oct;58(10):1729-1730. doi: 10.1111/jpc.16211. Epub 2022 Sep 13. No abstract available. PMID 36098673
- [Result] Genuis SJ, Lipp C. Ethical diversity and the role of conscience in clinical medicine. Int J Family Med. 2013;2013:587541. doi: 10.1155/2013/587541. Epub 2013 Dec 12. PMID 24455248
- [Result] Lehmann LS, Sulmasy LS, Desai S; ACP Ethics, Professionalism and Human Rights Committee. Hidden Curricula, Ethics, and Professionalism: Optimizing Clinical Learning Environments in Becoming and Being a Physician: A Position Paper of the American College of Physicians. Ann Intern Med. 2018 Apr 3;168(7):506-508. doi: 10.7326/M17-2058. Epub 2018 Feb 27. PMID 29482210
- [Result] Beran TN, Altabbaa G, Oddone Paolucci E. Observational Study of Conformity in Yet Another Medical Learning Environment: Conformity to Preceptors During High-Fidelity Simulation. Adv Med Educ Pract. 2023 Dec 22;14:1445-1452. doi: 10.2147/AMEP.S427996. eCollection 2023. PMID 38149121
- [Result] Beran TN, McLaughlin K, Al Ansari A, Kassam A. Conformity of behaviors among medical students: impact on performance of knee arthrocentesis in simulation. Adv Health Sci Educ Theory Pract. 2013 Oct;18(4):589-96. doi: 10.1007/s10459-012-9397-5. Epub 2012 Aug 31. PMID 22936210
- [Result] Beran TN, Kaba A, Caird J, McLaughlin K. The good and bad of group conformity: a call for a new programme of research in medical education. Med Educ. 2014 Sep;48(9):851-9. doi: 10.1111/medu.12510. PMID 25113112